CLINICAL TRIAL: NCT05751746
Title: The Effect of Peripartum Magnesium Sulfate Use on the Occurrence of Postpartum Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-2209-780-302
Record Dates: First submitted 2023-01-30; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Control group with participants who do not get magnesium sulfate administration.
- Magnesium group: Intervention group with participants who get magnesium sulfate administration.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — Magnesium sulfate will be administered following a protocol that obstetricians already use in our hospital.
  Groups: Magnesium group

SUMMARY:
This is an observational study that will be conducted on pregnant women under vaginal delivery or cesarean section. The magnesium sulfate will be given to appropriate participants with a protocol that obstetrician are already using in our hospital. After delivery, participants are asked to answer sequential questionnaires to assess postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who will do delivery.
* Gestational week >= 30 week
* Singleton

Exclusion Criteria:

* History of depression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are all pregnant women.
Study Population: This is aimed adult singleton pregnant women with gestation age more than 30 weeks who are scheduled to give birth. Participants who get peripartum administration of magnesium sulfate are classified as magnesium group, and participants who do not get magnesium sulfate administration are classified as control group.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
postpartum depression | 6 week after discharge
  depression diagnosis using K-EPDS(Korean version of Edinburgh Postnatal Depression Scale) on a scale of 7 to 30 points.
postpartum depression severity | 6 week after discharge
  depression severity using K-EPDS; mild (7~13 points), moderate (14~19 points), severe (20~30 points)

SECONDARY OUTCOMES:
postpartum depression | 2week after discharge
  depression diagnosis using K-EPDS(Korean version of Edinburgh Postnatal Depression Scale) on a scale of 7 to 30 points.
postpartum depression severity | 2 week after discharge
  depression severity using K-EPDS; mild (7~13 points), moderate (14~19 points), severe (20~30 points)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonguido, South Korea

IPD SHARING:
Plan to Share IPD: No